CLINICAL TRIAL: NCT04533100
Title: The Association of Protein-Energy Adequacy With Mortality in Critically Ill Patients With Acute Kidney Injury. A Prospective Observational Single- Centre Study.
Brief Title: The Association of Protein-Energy Adequacy With Mortality in Critically Ill Patients With Acute Kidney Injury.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Mohd Shahnaz, MBBS, M Anes, Principal Investigator., University of Malaya
Other Study IDs: MREC ID NO: 2018222-6043
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Critical Illness; Acute Kidney Injury
Keywords: Protein; Energy; Adequacy; Mortality
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational single-center study in which the association of Protein-Energy Adequacy and 28-Days of Mortality among critically ill patients with Acute Kidney Injury, AKI will be investigated. The association of Protein-Energy adequacy with a length of ICU and hospital stay, total ventilator, and inotropic drug days among critically ill patients with AKI also will be investigated.

DETAILED DESCRIPTION:
Patients with Acute Kidney Injury, AKI are probably more exposed to the risk of malnutrition especially if they undergo Renal Replacement Therapy, RRT. Optimization of nutrients especially energy and protein can ensure a better health outcome for critically ill patients with AKI. Moreover, there is no research on the association of Protein- Energy adequacy with mortality among critically ill patients with AKI in Malaysia. So, the main purpose of this study is to investigate the relationship of Protein-Energy adequacy with mortality among critically ill patients with AKI

Subjects will be recruited upon admission in ICU after fulfilling the inclusion and exclusion criteria. They will be follow up from day 1 until day 14 or until ICU Discharge. Data including Demographic, Clinical, Laboratory, and Nutritional Status will be recorded. On Day 28, the outcome data including Mortality, length of ICU Stay, and Length of Ventilator day will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years old and older
2. Patients who are admitted to the participating ICU.
3. Patients who are mechanically ventilated.

Exclusion Criteria:

1. Patients who are less than 18 years old
2. End-stage renal disease patients
3. Patients undergo kidney transplantation within 3 months before ICU admission
4. Pregnant patients
5. The patient is moribund with expected death within 24 hour or whom survival to 28 days is unlikely due to uncontrollable comorbidity (cardiac, pulmonary or hepatic end-stage disease; hepatorenal syndrome; poorly controlled cancer; severe post-anoxic encephalopathy and others)
6. Prior treatment with RRT within 30 days
7. Anticipated alive ICU discharge within 24 hours
8. Readmission to the ICU during the same hospitalization episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in adult Intensive Care Unit, University Malaya Medical Centre (UMMC), Malaysia.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
28-Days Mortality | 1 day
  Mortality status of subjects on day 28 from recruitment.

SECONDARY OUTCOMES:
Length of ICU Stay | 1 day
  Duration of ICU Stay from ICU admission until ICU discharge
Length of Ventilator Day | 1 day
  Duration of ventilator used by subjects from ICU admission until ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: MOHD SHAHNAZ HASAN, MBBS, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: ESPEN Guideline on Clinical Nutrition in the Intensive Care Unit. Clinical Nutrition — https://doi.org/10.1016/j.clnu.2018.08.037